CLINICAL TRIAL: NCT03200002
Title: Effect of Cyclophosphamide Versus Mycophenolate Mofetil in Induction Therapy of Lupus Nephritis in Nepalese Population
Brief Title: Cyclophosphamide Versus Mycophenolate Mofetil in Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chitwan Medical College (Other)
Responsible Party: Principal Investigator, Arun Sedhain, Associate Professor, Chitwan Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LN_CYC_MMF
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: To Compare the Effects of Mycophenolate Mofetil With Cyclophosphamide in Neplaese Lupus Nephritis Patients
Keywords: Lupus Nephritis, cyclophosphamide, Mycophenolate mofetil
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclophosphamide (Experimental): Participants in this arm received intravenous cyclophosphamide (CYC) in the dose of 0.5 to 1 gram per m2 of body surface area.
  Interventions: Drug: Cyclophosphamide
- mycophenolate mofetil (Experimental): Patients in this arm received mycophenolate mofetil in the tablet form.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide injection was administered in the dose of 0.5 to 1 gram per m2 of body surface area. The medicine, which is available in the strength of 1 gram in powder form, was first dissolved in 20 ml of normal saline. Only15 ml of this preparation was mixed in 100 ml of normal saline and was infused over a period of one hour. CYC was not given to those patients who had total leukocyte counts (TLC) less than 2500/mm3. Those patients were re-evaluated after one week and intravenous pulse CYC was reinstituted if the TLC exceeds 2500/mm3. Pulse CYC was administered every month for a total of six infusions.
  Arms: Cyclophosphamide
Drug: Mycophenolate Mofetil — Participants in the MMF group were administered tablet mycophenolate mofetil at a starting dose of 500 mg twice daily if the weight of the patient was less than 50 kilograms and 750 mg twice daily if the weight was more than 50 kilograms. After one month, the dose of MMF was increased to 750 mg twice daily. The clinical response was monitored in terms of reduction in serum creatinine and proteinuria. MMF dose was decreased or interrupted in patients experiencing an absolute neutrophil count <1300/mm3 at any study visit; MMF treatment was discontinued if a patient experienced an absolute neutrophil count <1000/mm3.
  Arms: mycophenolate mofetil

SUMMARY:
This was a prospective open label randomized control trial, which was conducted for a period of one and half year from January 2014 to June 2015. Out of 52 patients screened, 49 patients meeting the international society of nephrology/ renal pathology society (ISN/RPS) criteria were enrolled in the study comprising of 25 and 24 patients in the cyclophosphamide (CYC) and mycophenolate mofetil (MMF) groups respectively. Forty two patients (21 in each group) could complete the study till the end of 6 months and were included in final analysis. Baseline clinical evaluation and investigations were done and recorded. CYC was given intravenously as a monthly pulse in the dose of 0.5 to 1 gram per m2 body surface area. MMF was administered in the tablet form with the starting dose of 500 mg twice daily, which was increased to 750 mg twice daily after a month. Patients were assessed and monitored monthly and the details were recorded. Efficacy of treatment was measured as primary end point for those who achieved partial remission (reduction of 24 hour urinary protein to < 3.5gms/day if baseline proteinuria >3.5 gms/day or decrease by 50% if baseline proteinuria <3.5 gms/day) and secondary end point for those who achieved complete remission (normalization of serum creatinine and < 500 mg of 24 hour urinary protein). Adverse events experienced by the patients were also recorded during monthly visit.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease associated with multiple organ involvement, among which kidney involvement, also known as lupus nephritis (LN), is quite common in SLE. LN is associated with a more than four-fold increase in mortality in patients with SLE. The management of SLE and LN comprises timely and coordinated management consisting of initial or induction phase of aggressive immunosuppression to bring the active disease under control followed by maintenance phase. The initial phase usually lasting for six months consists of treatment with steroid and cyclophosphamide or mycophenolate mofetil. So far there is no study published regarding the efficacy and adverse events of such treatments in Nepal. So, this study aimed to evaluate and compare the effectiveness and safety profile of mycophenolate mofetil and intravenous pulse cyclophosphamide in induction therapy of LN in Nepalese population.

A total of 52 patients with international society of Nephrology/ renal pathology society (ISN/RPS) class III to V lupus nephritis were screened, 3 of which did not meet entry criteria and 49 patients were enrolled in the study comprising of 25 and 24 patients in the MMF and CYC group respectively. Twenty one patients in each groups could complete the study till the end of 6 months and were included for analysis.

Patients in the CYC group received intravenous cyclophosphamide (CYC) in the dose of 0.5 to 1 gram per m2 of body surface area. The medicine, which is available in the strength of 1 gram in powder form, was first dissolved in 20 ml of normal saline. Only15 ml of this preparation was mixed in 100 ml of normal saline and was infused over a period of one hour. CYC was not given to those patients who had total leukocyte counts (TLC) less than 2500/mm3. Those patients were re-evaluated after one week and intravenous pulse CYC was reinstituted if the total leucocyte count (TLC) exceeds 2500/mm3. Pulse CYC was administered every month for a total of six infusions.Patients were monitored monthly and the details were recorded. During follow ups, any adverse events in between were noted and detailed physical evaluation was done and all baseline investigations (except USG abdomen, chest X-ray, serum anti nuclear antibody (ANA) and anti double strain deoxy-ribonuccleic acid (anti dsDNA), complement factor 3 (C3) and complement facotr 4 (C4) level) was repeated. Fasting lipid profile was repeated at the end of third and sixth month of treatment.

During the course of treatment, if a patient had interruption of medication for less than a 10 days' period due to any reason, s/he was considered as a regularly included subject. If the interruption extended beyond 10 days, the patient was withdrawn from the study.

Patients in the MMF group were administered tablet mycophenolate mofetil at a starting dose of 500 mg twice daily if the weight of the patient was less than 50 kilograms and 750 mg twice daily if the weight was more than 50 kilograms. After one month, the dose of MMF was increased to 750 mg twice daily. The clinical response was monitored in terms of reduction in serum creatinine and proteinuria. MMF dose was decreased or interrupted in patients experiencing an absolute neutrophil count <1300/mm3 at any study visit; MMF treatment was discontinued if a patient experienced an absolute neutrophil count <1000/mm3.

All patients, irrespective of randomized group, received concomitant corticosteroid therapy with oral prednisolone and hydroxychloroquine. Angiotensin receptor inhibitors (ACEi)/ angiotensin receptor blocker (ARBs) were given to all patients if the blood pressure remained above or equal to 120 mmHg of systolic blood pressure and 80 mmHg of diastolic blood pressure. If the blood pressure remained persistently high despite the use of ACEi/ARBs, other antihypertensives were added as required to achieve target blood pressure <130/80 mmHg. Oral prednisolone was given at an initial dose of 1 mg/kg with a maximum dose of 60 mg/day. The starting dose of prednisolone was continued for initial one month. Then, the dose of oral prednisolone was tapered at the rate of 10 mg/day every 2 weeks and was maintained at the baseline dose of 5 to 7.5 mg per day then after. Additional intravenous methylprednisolone was given at the beginning of treatment for patients who presented as rapidly progressive glomerulonephritis (RPGN) and who had activity index of more than 8 out of 24 on kidney biopsy irrespective of the randomized group (MMF or CYC) of the patient. The dose of methylprednisolone was 1 gram, which was given after mixing with 100 ml of normal saline and was infused intravenously over 1 hour for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed LN with ISN/RPS histopathology classes III to V

Exclusion Criteria:

* Patients with biopsy had proven ISN / RPS classes I, II and VI LN
* Patients with previous history of treatment and relapse of lupus nephritis
* Patients who were receiving continuous dialysis for more than two weeks prior to randomization.
* Patients of less than 12 years of age
* Patients who had concurrent infection or illness at the time of enrollment
* Patients who were taking concurrent medications which are supposed to have interactions with MMF or CYC
* Female patients who were pregnant and breastfeeding.
* Patients who did not give consent for participation

Ages: 13 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
partial remission | 6 months
  reduction of 24 hour urinary protein to < 3.5gms/day if baseline proteinuria >3.5 gms/day or decrease by 50% if baseline proteinuria <3.5 gms/day

SECONDARY OUTCOMES:
Complete remission | 6 months
  normalization of serum creatinine and < 500 mg of 24 hour urinary protein

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sedhain A, Hada R, Agrawal RK, Bhattarai GR, Baral A. Low dose mycophenolate mofetil versus cyclophosphamide in the induction therapy of lupus nephritis in Nepalese population: a randomized control trial. BMC Nephrol. 2018 Jul 11;19(1):175. doi: 10.1186/s12882-018-0973-7. PMID 29996800